CLINICAL TRIAL: NCT01533324
Title: Phase II Study of S-1 Combined With Calcium Folinate to Treat Advanced Hepatocellular Carcinoma
Brief Title: S-1/LV One Week on and One Week Off Regimen in Advanced Hepatocellular Carcinoma (HCC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Military Medical University (Other)
Responsible Party: Principal Investigator, Xie feng, attending physician, Second Military Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC-SL-2W
Record Dates: First submitted 2012-02-10; First posted 2012-02-15 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Carcinoma; Liver Diseases; Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; S-1; Leucovorin; fluorouracil
MeSH Terms: conditions — Carcinoma; Liver Diseases; Carcinoma, Hepatocellular | interventions — Leucovorin; titanium silicide; Formyltetrahydrofolates

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- S-1 combined with LV (Experimental): S-1 combined with LV
  Interventions: Drug: S-1 combined with Leucovorin

INTERVENTIONS:
Drug: S-1 combined with Leucovorin — S-1 capsules 80mg/m2/d BID one week on and one week off Leucovorin tablets 50mg/d BID one week on and one week off
  Other Names: TS-1; formyltetrahydrofolate

SUMMARY:
S-1 is a new chemotherapy drug. Some phase II trials showed S-1 is effective in Hepatocellular Carcinoma (HCC). S-1 combined with calcium folinate (SL) showed very good efficiency and safety in colorectal cancer (CRC). The short duration (two weekly regimen) is better than common course 4 week regimen in tolerance. So the investigators want to examine the efficiency and safety of SL one week on and one week off regimen in HCC.

DETAILED DESCRIPTION:
S-1 is a new chemotherapy drug. Some phase II trials showed S-1 is effective in HCC. S-1 combined with calcium folinate (SL) showed very good efficiency and safety in CRC. The short duration (two weekly regimen) is better than common course 4 week regimen in tolerance. So the investigators want to examine the efficiency and safety of SL one week on and one week off regimen in HCC.

SL one week on and one week off regimen will be give to advanced HCC patients. The primary endpoint is durable complete response (DCR).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 70 years > Age > 18 years
* Patient with unresectable primary hepatocellular carcinoma
* Child-Pugh Class A or B, without ascites
* ECOG score 0
* At least one tumor nodule can be evaluated by CT or MRI
* Can take medicine orally
* Expected survival time not less than 12 weeks
* Women of childbearing potential must have a negative pregnancy test performed within 7 days prior to enrolling in this portion of the study During the trial and 4 week after the trial, must take contraception
* Patients must be:
* Hemoglobin > 9.0g/dl
* ANC > 1.5×109/L
* Platelet ≥ 60×109/L
* Total bilirubin < 3mg/dl
* ALT or AST < 5 X ULN
* ALP < 4 X ULN
* PT-INR < 2.3
* Patients who is taking Warfarin , should be tested every week till getting stable INR
* Serum creatinine < 1.5 X ULN
* Serum amylase and lipase < 2 X ULN

Exclusion Criteria:

* Known or suspected allergy to any agent given in association with this trial
* Local treatment within 4 weeks prior to start of study drug
* History of any heart disease
* History of HIV infection except for HBV and HCV
* Active clinically serious infections (> 2 NCI-CTC Version 3.0)
* Clinically significant gastrointestinal bleeding within 4 weeks prior to study entry.
* Embolization or infarction such as transient ischemic disease, deep vein thrombosis, pulmonary embolization within 6 months prior to study entry
* Previous malignancy (except for cervical carcinoma in situ, adequate treated basal cell carcinoma, or superficial bladder tumors [Ta, Tis and T1], early gastric cancer, or other malignancies curatively treated > 3 years prior to entry
* Extrahepatic tumor spread which affects patient's prognosis, such as bony metastasis or brain metastasis
* Hydrothorax， ascites and hydropericardium need to drain
* Serious diarrhea
* Combined with serious pulmonary diseases, such as interstitial pneumonia, pulmonary fibrosis and serious pulmonary emphysema
* Serious complication,such as intestinal obstruction,renal insufficiency, hepatic insufficiency and cerebrovascular disorders
* Pregnant or breast-feeding
* Any condition that is unstable or could jeopardize the safety of the patient and its compliance in the study, in the investigator's judgment.
* Gastrointestinal disease that may affect to the absorption of drug or pharmacokinetics.
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in this study
* Patients unable to swallow oral medications.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2011-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
DCR | in two years
  DCR means patient got the best reaction and last for more than 4 weeks DCR=（CR）+ （PR）+ （SD） by RESIST 1.1

SECONDARY OUTCOMES:
TTP ( time to progression) | in 2 years
  from enrolled to progression(iconography).
OS ( overall survival) | in two years
  to death
safety | in two years
  any adverse reaction by NCI-CTCAE 3.0

CONTACTS AND LOCATIONS:
Overall Officials: Yang Jiamei, Chief, Study Chair — Second Military Medical University
Locations (1):
- Eastern Hepatobiliary Surgery Hospital, Shanghai, Shanghai Municipality, China